CLINICAL TRIAL: NCT05809934
Title: A Randomised, Double-blind, Placebo-controlled, Multi-centre Phase 2b Study to Evaluate the Efficacy, Safety and Tolerability of AZD2693 in Participants With Non-cirrhotic Non-alcoholic Steatohepatitis (NASH) With Fibrosis Who Are Carriers of the PNPLA3 rs738409 148M Risk Allele
Brief Title: A Study to Evaluate AZD2693 in Participants Who Are Carriers of the PNPLA3 148M Risk Allele With Non-cirrhotic Non-alcoholic Steatohepatitis With Fibrosis
Acronym: FORTUNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7830C00004; 2023-509704-14-00 (Registry Identifier: CTIS (EU)); 2022-001629-65 (EudraCT Number)
Record Dates: First submitted 2023-02-23; First posted 2023-04-12 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Steatohepatitis; NASH; fatty liver disease; Non alcoholic fatty liver; liver fibrosis; PNPLA3 148M Risk Allele; Non Cirrhotic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: Randomised, Double-blind, Placebo-controlled, Multi-centre Phase 2b Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AZD2693 dose 1 (Experimental): Participants will receive AZD2693 dose 1
  Interventions: Drug: AZD2693
- AZD2693 dose 2 (Experimental): Participants will receive AZD2693 dose 2
  Interventions: Drug: AZD2693
- Placebo (Placebo Comparator): Participants in this arm will receive placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AZD2693 — AZD2693 solution SC once per month
  Arms: AZD2693 dose 1; AZD2693 dose 2
Other: Placebo — Sodium chloride 0.9% solution SC once per month
  Arms: Placebo

SUMMARY:
A Study to Evaluate the Efficacy, Safety and Tolerability of AZD2693 given by subcutaneous injection in adult participants with non-cirrhotic non-alcoholic steatohepatitis with fibrosis and who are carriers of the PNPLA3 148M Risk Allele

ELIGIBILITY:
Key Inclusion Criteria :

Participants are eligible to be included in the study only if all the following criteria apply:

Age

1. Participant must be 18 to 75 years of age (inclusive) at the time of signing the informed consent.

   Type of Participant and Disease Characteristics
2. Participants who are carriers for the PNPLA3 rs738409 148M risk allele.
3. Participants with histological evidence of NASH based on central pathologist evaluation of a liver biopsy obtained up to 6 months before randomisation, or during screening, fulfilling both criteria:

   1. Definitive NASH with NAS ≥ 4 with ≥ 1 in each component (ie, steatosis, lobular inflammation, and ballooning).

   <!-- -->

   1. Presence of fibrosis stage F2 or F3 according to the NASH CRN fibrosis staging system based on central pathologist evaluation.

Key Exclusion Criteria :

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Liver disease of other aetiologies (eg, alcoholic steatohepatitis; drug-induced, viral or autoimmune hepatitis; primary biliary cirrhosis; primary sclerosing cholangitis; hemochromatosis; alpha-1 antitrypsin deficiency; Wilson's disease)
2. History of cirrhosis and/or hepatic decompensation, including ascites, hepatic encephalopathy, or variceal bleeding.
3. Historical persistent or pre-existing renal disease marked by eGFR < 40 mL/min/1.73 m2 (as defined by Kidney Disease Improving Global Outcomes guidelines).
4. Confirmed platelet count outside the normal range at the screening visit.
5. Any of the following confirmed at the screening visit:

   1. ALT > 5.0 × ULN
   2. TBL > 1.5 mg/dL (TBL > 1.5 mg/dL is allowed if conjugated bilirubin is < 1.5 × ULN)
   3. INR > 1.3
   4. ALP > 1.5 × ULN (unless the ALP elevation is not from hepatic origin as determined by a bone-specific ALP)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2025-07-14 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving NASH resolution without worsening of fibrosis based on histology after 52 weeks treatment | after 52 weeks
  To assess the effect of AZD2693 versus placebo on histological resolution of NASH in participants with non-cirrhotic NASH with fibrosis and PNPLA3 risk allele carriers after 52 weeks

SECONDARY OUTCOMES:
Proportion of participants with at least one stage of liver fibrosis improvement with no worsening of NASH based on biopsy after 52 weeks treatment | after 52 weeks
  To assess the effects of AZD2693 versus placebo on histological fibrosis improvement
Proportion of participants with ≥ 2-point improvement from baseline in NAS based on biopsy after 52 weeks treatment | after 52 weeks
  To assess the effect of AZD2693 versus placebo on ≥ 2-point improvement in NAS
Proportion of participants with improvement in fibrosis by at least one stage based on biopsy after 52 weeks treatment | after 52 weeks
  To assess the effect of AZD2693 versus placebo on improvement in fibrosis by at least one stage

OTHER OUTCOMES:
Number of participants with Adverse Events/Serious Adverse Events (AEs/SAEs) and abnormal laboratory test results | 64 weeks
  Haematology, urinalysis, clinical chemistry and eGFR
Number of participants with Adverse Events/Serious Adverse Events (AEs/SAEs) and abnormal clinical test results | 64 weeks
  Vital signs and electrocardiogram (ECG) assessments

CONTACTS AND LOCATIONS:
Locations (141):
- United States (36):
  - Research Site, Chandler, Arizona
  - Research Site, Peoria, Arizona
  - Research Site, Surprise, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Gardena, California
  - Research Site, La Mesa, California
  - Research Site, Lancaster, California
  - Research Site, Los Angeles, California
  - Research Site, Montclair, California
  - Research Site, Orange, California
  - Research Site, Rialto, California
  - Research Site, Santa Ana, California
  - Research Site, Boca Raton, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Marietta, Georgia
  - Research Site, Topeka, Kansas
  - Research Site, Detroit, Michigan
  - Research Site, Las Vegas, Nevada
  - Research Site, Westlake, Ohio
  - Research Site, Chickasha, Oklahoma
  - Research Site, Hershey, Pennsylvania
  - Research Site, Summerville, South Carolina
  - Research Site, Cordova, Tennessee
  - Research Site, Austin, Texas
  - Research Site, Brownsville, Texas
  - Research Site, Denison, Texas
  - Research Site, Edinburg, Texas
  - Research Site, Houston, Texas
  - Research Site, Red Oak, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Seattle, Washington
- Argentina (6):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, La Plata
  - Research Site, Mar del Plata
  - Research Site, San Juan Bautista
- Brazil (5):
  - Research Site, Botucatu
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Chile (2):
  - Research Site, Santiago
  - Research Site, Valdivia
- China (16):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Liaocheng
  - Research Site, Nanchang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Wenzhou
  - Research Site, Xi'an
  - Research Site, Xuzhou
  - Research Site, Zhenjiang
- Research Site, Cartagena, Colombia
- Germany (4):
  - Research Site, Konstanz
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, Münster
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- India (4):
  - Research Site, Hyderabad
  - Research Site, Jaipur
  - Research Site, Punjab
  - Research Site, Surat
- Italy (5):
  - Research Site, Milan
  - Research Site, Palermo
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Torino
- Japan (22):
  - Research Site, Bunkyō City
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Gifu
  - Research Site, Kagoshima
  - Research Site, Kawasaki-shi
  - Research Site, Kobe
  - Research Site, Kumamoto
  - Research Site, Kure-shi
  - Research Site, Kurume-shi
  - Research Site, Kyoto
  - Research Site, Minatoku
  - Research Site, Nagoya
  - Research Site, Okayama
  - Research Site, Omura-shi
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Shinjuku-ku
  - Research Site, Takasaki-shi
  - Research Site, Tsu
  - Research Site, Yokohama
- Malaysia (4):
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Pulau Pinang
  - Research Site, Seremban
- Mexico (6):
  - Research Site, Acapulco
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, Torreón
  - Research Site, Veracruz
  - Research Site, Xalapa
- Peru (2):
  - Research Site, Chorrillos
  - Research Site, Lima
- Philippines (4):
  - Research Site, Cebu
  - Research Site, Puerto Princesa City
  - Research Site, Roxas City
  - Research Site, San Fernando City
- Research Site, Singapore, Singapore
- South Korea (2):
  - Research Site, Junggu
  - Research Site, Seoul
- Spain (5):
  - Research Site, A Coruña
  - Research Site, Almería
  - Research Site, Lleida
  - Research Site, Málaga
  - Research Site, Zaragoza
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
- Turkey (Türkiye) (6):
  - Research Site, Adana
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Eskişehir
  - Research Site, Izmir
  - Research Site, Rize
- Research Site, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home